CLINICAL TRIAL: NCT02723266
Title: Supporting American Indian/Alaska Native Mothers and Daughters in Reducing Gestational Diabetes Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Colorado, Denver (Other); University of Oklahoma (Other); Sundance Research Institute (Unknown); St. Regis Mohawk (Unknown); Indian Health Care Resource Center of Tulsa (Unknown); Children's Hospital of Philadelphia (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Denise Charron-Prochownik, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01NR014831-01A1 (NIH)
Record Dates: First submitted 2016-03-01; First posted 2016-03-30 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Gestational Diabetes Mellitus
Keywords: American Indian, Alaska Native Adolescents; Preconception Counseling; Reproductive Health; Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Treatment receives the STOPPING-GDM intervention. Control does not receive the intervention.
  Interventions: Behavioral: STOPPING-GDM
- Control (No Intervention): Control does not receive the intervention.

INTERVENTIONS:
Behavioral: STOPPING-GDM — Educational counseling and skills building Intervention
  Arms: Intervention

SUMMARY:
The purpose of this study is to modify an existing Reproductive Health intervention for adolescents with diabetes for Gestational Diabetes and make it culturally appropriate American Indian/Alaska Native adolescents. The intervention will then be evaluated for effectiveness in AI/AN female teens at risk for GDM.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) has escalated to epidemic proportion and can cause maternal and child complications. GDM is a significant maternal risk factor for subsequent development of type 2 diabetes (T2D) and places the fetus at increased risk for congenital morbidity/mortality and for future onset of diabetes. American Indian and Alaska Native (AI/AN) women are twice as likely to develop GDM and T2D; mostly due to healthcare disparities (e.g., limited access to resources, lack of culturally relevant programs). The need for an inexpensive accessible GDM intervention in this population is compelling. The intervention should be delivered during adolescence and prior to sexual debut. Preconception counseling (PC) prevents unplanned pregnancies and significantly reduces risks of complications. If GDM in a previous pregnancy is an indicator of high risk in subsequent pregnancies, then preventing GDM in a first pregnancy is imperative. For a significant and innovative shift in paradigm, the Investigators propose a primary prevention PC intervention for AI/AN adolescent females at risk for GDM to enhance healthy lifestyle behaviors and family planning vigilance prior to this first pregnancy. The Investigators will target girls starting at the age of 12 to coincide with both the "Coming-of-Age" rituals for AI/AN girls during which many receive womanly advice from elder female family members, and the American Diabetes Association recommendation that PC in all females should start at puberty. This new directive will require support from the teens' mothers (or their female caregiver) and well-informed community health care professionals (HCP). Our objective is to adapt our current PC intervention (validated for teens with diabetes) using a sequential mixed-method design with a multi-tribal AI/AN community-based participatory research (CBPR) approach (e.g., Navajo, Cherokee, 40 Oklahoma tribes; 8 project members are AI/AN) by first using focus groups of teens, mothers, HCP, and Tribal leaders; and then testing this culturally appropriate PC theory-based intervention named Stopping GDM in AI/AN adolescent females 12 to <20yrs at risk for GDM (e.g., pre-diabetes or BMI> 85%). Teens and their mothers will receive the Stopping GDM to raise their awareness of the risks of GDM and benefits of healthy lifestyle to reduce these risks. By also providing mothers with PC knowledge and skills they can naturally weave cultural/social influences into their communications with their daughters. The multi-level intervention will be directed at the individual, familial and institutional levels simultaneously. AI/AN community-researcher partnerships have been established. A randomized controlled trial with a 15mos follow-up will test the effects of receiving online Stopping GDM on mother-daughter (M-D) cognitive/psychosocial and behavioral outcomes, and daughter family planning vigilance. The final online Stopping GDM program will be provided at no cost to the Indian Health Service (IHS) for dissemination to all their sites. HCPs at each clinical facility will be given free access to a continuing education program for PC training. This proposal provides a unique opportunity for a broad dissemination to significantly impact all IHS AI/AN female teens at risk for GDM, and help to prevent them and their future children from developing T2D.

ELIGIBILITY:
Inclusion Criteria: Daughter(index subject)

* females between the ages of 12 to <20 years
* at risk for GDM (such as having metabolic syndrome, pre-diabetes, or BMI > 85%; and an A1C < 6.5%)
* fluent in English.

Inclusion criteria: Mother (or significant female caregiver, e.g., grandmother, aunt, adult sister, stepmother) of daughters at risk for GDM

* natural, adoptive, or step, living with their daughters
* fluent in English

Exclusion Criteria: Daughters:

* A1C > 6.5%, [20, 26] abnormal Glucose Tolerance Test (GTT),
* signs and symptoms of diabetes,
* a history of another chronic illness or mental retardation,
* pregnant at the time of recruitment.

Exclusion Criteria Mothers:

* foster mother of an adolescent girl because she may not be a consistent caregiver.

Ages: 12 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 398 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Reproductive Health Behaviors | 15 months
  Family-Planning Vigilance Behavior are defined as using effective family planning/abstinence, seeking PC, and initiating discussion with health care professionals . "Effective family planning behaviors" is a weight summary of the teen's most frequently used contraception. Weights will be derived using the annual failure rates for methods of contraception reported in Trussell's algorithm. Rates are transformed into probabilities of failure (0 to 1), 0 = no failure. Overall effectiveness of contraception is computed as 1-Pr [Failure]. Combination methods (> 2 jointly) is the product of the failure probability of the individual methods used jointly. For multiple methods used singly, the overall probability of failure will be computed as the average of the failure probabilities. Subjects who were never sexually active will be given a failure probability of zero
Beliefs and Attitudes | 15 months
  Beliefs/attitudes Reproductive Health and Diabetes Questionnaire (EHBM scale) Based on the EHBM,[53, 76, 82] perceived susceptibility (9 items) and perceived severity (7), perceived benefits (12) of and barriers (15), and self-efficacy (18) (confidence to use FPV); Likert-type (1=strongly disagree to 7=strongly agree).[76] Each construct has a composite score; higher= stronger attitudes. (alphas: susceptibility = .74; severity = .94; benefit = .88; barriers = .97; self-efficacy = .96
Knowledge/Decision-Making | 15 Months
  Knowledge/decision-making Reproductive-health Awareness for Teens with DM Quest (Knowledge scale) Multiple choice, based on 100% correctness, subscales: diabetes and pregnancy (28 items); contraception (5); sexuality (7); puberty (3); PC (25); and general family planning (8) (Cronbach alpha .71; test-retest reliability r= 0.76). Split-half differentiates pre- from post-test
Social Support | 15 months
  Social Support Reproductive Health and Diabetes Q. (Social Support scale) Social support is the process by which help is obtained from the social network (e.g., mothers/ female guardian) to meet one's needs. Support measure for mothers is the perceived actual support (emotional, appraisal, informational, and instrumental)[54] they provided to their daughters for lifestyle management and family planning vigilance. Daughters' measure is perceived available support from their mother for the same behaviors. Summation score of 9 items with responses, "a lot of help" =7 to "no help at all" =1. Higher scores = greater support. Alpha = .92
Initiating Discussion | 15 months
  Initiating Discussions with M-D Initiating Discussion M-D Scale Teens and mothers respond to 4 yes/no items of actual discussions they have had regarding GDM and reproductive health issues (pregnancy, sexuality, birth control and PC
Lifestyle Management | 15 months
  Lifestyle Self-Management Lifestyle Self-Management Scale (DM Care Profile) Daughter's adherence is a 3-item scale (1= "not very well done" to 7= "very well done") based on diabetes-prevention self-care management (diet, physical activity, clinic visits).[84] Cronbach's alpha from our studies is .75. Culturally-relevant items will be added during Phase 1

SECONDARY OUTCOMES:
BMI | 15 months
  Body Mass Index (BMI) BMI percentile a standard parameter for obesity will be the measured weight (kilograms) divided by measured height using a stadiometer (meters) squared. Change in BMI will be analyzed. Percentiles will be specific to sex and month of age using algorithms by the Center for Disease Control. BMI z scores will also be calculated. Identical scales and stadiometers, provided by the study, will be calibrated according to the manufacturer. Protocols/ categories from the SEARCH study will be used.
Hemoglobin A1C values to evaluate Glycemic Control | 15 months
  Glycosylated Hemoglobin (A1C) A1C is a standard index of long-term glycemic control, reflecting 3-month average blood glucose levels. Clinic A1C values will be recorded from the subjects' medical records, and entered into the online database. Each site uses the same standardized method for obtaining A1C samples. Blood will be collected from a finger stick and analyzed immediately. Each site will use the same manufacturer's calibration techniques . The investigators will evaluate changes in glycemic control per the categories in the American Diabetes Association guidelines. A Glycosylated Hemoglobin (A1C) > 6.5% is an exclusion criteria.
Number of subjects reporting an unplanned pregnancy | 15 months
  Self Report of Unplanned Pregnancy (no or yes) since last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy O'Bannion, MS, Study Director — Indian Health Care Resource Center of Tulsa; Jeff Powell, MD, Study Director — University of Colorado (Shiprock-subcontract )
Locations (1):
- Indian Health Resource Center of Tulsa, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
It is our intention to make all data generated from this proposal freely available. The primary mechanism of data dissemination will be through submission of abstracts to regional, national, and international meetings and the submission of manuscripts. The principal investigator will serve as liaison with other investigators in the sharing of additional materials if necessary.